CLINICAL TRIAL: NCT01822158
Title: Vaginal Delivery Debrief: A Nursing Research Study
Brief Title: Vaginal Delivery Debrief Checklist to Improve Team Communication
Acronym: VDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHS PSPH N 002
Record Dates: First submitted 2013-03-20; First posted 2013-04-02 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Other Specified Complications of Labor and Delivery
Keywords: Vaginal Delivery; Debrief; Medical Team Communication; Obstetrical Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaginal delivery debrief checklist (Other): Utilization of a Vaginal Delivery Debrief Checklist after vaginal deliveries for a period of three months, by team members who have consented to be a part of this study and who are present at vaginal deliveries. The Vaginal Delivery Debrief checklist consists of 2 levels. The first level includes a list of 6 key elements, such as APGAR scores,estimated blood loss, perineal repair, etc. The second level,or extended debrief, occurs whenever unanticipated outcomes, such as low APGAR scores, postpartum hemorrhage or a difficult delivery occurs. Team members complete the checklist after each delivery they attend.
  Interventions: Other: Vaginal Delivery Debrief Checklist

INTERVENTIONS:
Other: Vaginal Delivery Debrief Checklist — Participating team members will utilize Vaginal Delivery Debrief checklist

SUMMARY:
This study is to determine if using a standardized debrief checklist after vaginal delivery improves communication between the vaginal delivery health care team members and if using the checklist increases a sense of enhanced communication between team members.

DETAILED DESCRIPTION:
This is a study for providers who are a part of the health care team involved with vaginal delivery of newborns. A checklist has been developed that may improve communication between team members following birth. The goal of this study is to evaluate whether the checklist improves or enhances team member communication.

ELIGIBILITY:
Inclusion Criteria:

* Registered Nurses (RNs) and Licensed Practical Nurses (LPNs) in the Women's and Children's Services Department who attend vaginal deliveries as well as providers who attend vaginal deliveries at Providence St Peter Hospital Family Birth Center in Olympia Washington (WA).

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05-12 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Determine if there is a change in satisfaction with team communication following the use of a structured debrief checklist after vaginal deliveries. | Within 6 months of data collection
  An electronic opinion survey will be administered to participants both pre and post checklist utilization. The survey was derived from communication literature on medical teams such as the collaboration items and 3 subscales from the labour and delivery version of the Safety Attitudes Questionnaire (SAQ) and the Agency for Healthcare Research and Quality (AHRQ) TeamSTEPPS training program for high functioning medical teams.

SECONDARY OUTCOMES:
Determine if the use of a vaginal delivery debrief checklist will reduce documentation of conflicting data in the electronic medical record. | Within 6 months of data collection
  Utilizing the pre-validated Vaginal Delivery Debrief Medical Record Audit Tool, records will be examined pre and post use of the Vaginal Delivery Debrief Checklist. Assessment will be made to determine if there are fewer conflicting data points in the electronic medical record (EMR) for key elements following use of the Vaginal Delivery Debrief Checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Daren B Sachet, RN, BSN, MPA, Principal Investigator — Providence Health & Services
Locations (1):
- Providence St Peter Hospital 413 Lilly RD NE, Olympia, Washington, United States

IPD SHARING:
Plan to Share IPD: No